CLINICAL TRIAL: NCT03188393
Title: A Phase II Trial Assessing the Accuracy of Tumor Bed Biopsies in Predicting Pathologic Response in Patients With Clinical/Radiologic Complete Response After Neoadjuvant Chemotherapy in Order to Explore the Feasibility of Breast Conserving Treatment Without Surgery
Brief Title: Assessing the Accuracy of Tumor Biopsies After Chemotherapy to Determine if Patients Can Avoid Breast Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NRG Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: NRG-BR005; NCI-2016-01825 (Registry Identifier: CTRP); NRG-BR005; NRG-BR005 (Other: NRG Oncology); NRG-BR005 (Other: CTEP); U10CA180868 (NIH)
Record Dates: First submitted 2017-06-13; First posted 2017-06-15 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Invasive Breast Carcinoma; Stage II Breast Cancer; Stage IIA Breast Cancer; Stage IIB Breast Cancer; Stage IIIA Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Diagnostic (biopsy of breast) (Experimental): After completion of neoadjuvant therapy, patients undergo stereotactic biopsy of breast tumor any time prior to breast conserving surgery. Patients then undergo breast conserving surgery as per standard of care. Patients may also undergo postoperative radiation therapy per standard of care or adjuvant therapy at the investigator's discretion.
  Interventions: Procedure: Biopsy of Breast

INTERVENTIONS:
Procedure: Biopsy of Breast — Undergo stereotactic biopsy
  Other Names: Breast Biopsy

SUMMARY:
This phase II trial studies how well biopsy of breast after chemotherapy works in predicting pathologic response in patients with stage II-IIIA breast cancer undergoing breast conserving surgery. Tumor tissue collected from biopsy before surgery may help to check if chemotherapy destroyed the breast cancer cells and may be compared to the tumor removed during surgery to check if they are the same.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the accuracy of post-neoadjuvant systemic therapy (NST) image-directed tumor bed biopsy for pathologic complete response (pCR), defined as resolution of both invasive disease and ductal carcinoma in situ (DCIS), in cases of clinical and radiologic complete response with trimodality imaging.

SECONDARY OBJECTIVES:

I. To collect axillary pathology results, surgical staging methods (sentinel lymph node biopsy and/or axillary lymph node dissection), and management (surgery and/or radiation) in order to determine axillary nodal response to neoadjuvant chemotherapy and its relationship to breast pCR.

II. To correlate imaging results with pathologic nodal status following neoadjuvant chemotherapy for future planning of axillary management in the next study.

III. To retrospectively assess the negative predictive value (NPV) of a trimodality imaging algorithm in combination with the tumor bed biopsy for predicting pCR.

IV. To collect all trimodality imaging data to determine which combination of the trimodality imaging best identifies the group achieving pCR.

V. To correlate the number of needle cores and tumor bed clip retrieval with the NPV of the tumor site biopsy.

VI. To determine the clinical, imaging, pathologic, and molecular tumor factors associated with the highest NPVs of post-NST tumor bed biopsies.

VII. To improve identification and selection of patients with breast and possible axillary pCR for future trial planning, routine biomarkers (estrogen receptor [ER], progesterone receptor [PR], HER2 neu, and Ki67) will be collected to allow comparison to image/clinical complete response (CR), and tumor bed biopsies.

OUTLINE:

After completion of neoadjuvant therapy, patients undergo stereotactic biopsy of breast tumor any time prior to breast conserving surgery. Patients then undergo breast conserving surgery as per standard of care. Patients may also undergo postoperative radiation therapy per standard of care or adjuvant therapy at the investigator's discretion.

ELIGIBILITY:
Inclusion Criteria:

* The patient must have signed and dated an Institutional Review Board (IRB)-approved consent form that conforms to federal and institutional guidelines
* The patient must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Patients must have had ER analysis performed on the primary breast tumor collected prior to neoadjuvant therapy according to current American Society of Clinical Oncology (ASCO)/College of American Pathologists (CAP) guideline recommendations for hormone receptor testing; if negative for ER, assessment of progesterone receptor (PgR) must also be performed according to current ASCO/CAP Guideline Recommendations for hormone receptor testing. Patients who have a primary tumor that is hormone receptor-positive or hormone receptor-negative are eligible.
* Patients must have had HER2 testing performed on the primary breast tumor collected prior to neoadjuvant chemotherapy according to the current ASCO/CAP guideline recommendations for human epidermal growth factor receptor 2 testing in breast cancer; patients who have a primary tumor that is HER2-positive, HER2-equivocal, or HER2-negative are eligible
* Patients must have had a biopsy marker placed within the tumor bed with imaging confirmation (preferably mammogram but ultrasound or magnetic resonance imaging [MRI] is acceptable) of marker placement prior to neoadjuvant chemotherapy
* Patients with operable focal or multifocal (T1-T3, stage II or III invasive ductal carcinoma [all receptor phenotypes]), and who have completed neoadjuvant chemotherapy with a clinical complete response (by clinical examination)
* Patients with synchronous bilateral breast cancer are eligible if at least one of the synchronous breast cancers has a cCR, and the side with a cCR meets criteria. (Patients with previous contralateral invasive breast cancer treated with anti-cancer therapy are eligible.)
* Patients must have achieved a complete or near complete radiologic tumor response on breast imaging with mammogram, ultrasound, and MRI during or after completion of appropriate neoadjuvant chemotherapy defined as:

  * Mammogram with malignant appearing calcification or mass ≤ 1 cm; or
  * Ultrasound with a hypoechoic area ≤ 2 cm; or
  * Breast MRI not demonstrating a residual mass with rapid rise and washout type III kinetics.
* At the time of consent, the patient's intent must be to undergo breast conserving therapy.
* Patient must be able to undergo stereotactic-vacuum-assisted breast biopsy with clip placement after completion of neoadjuvant chemotherapy. (The patient must be enrolled on the study before performing the post-neoadjuvant stereotactic-vacuum-assisted breast biopsy.)
* Patient must have completed neoadjuvant chemotherapy.
* Patients with HER2-positive tumors must have received neoadjuvant anti-HER2 therapy (either with all or with a portion of the neoadjuvant chemotherapy regimen), unless medically contraindicated.
* Patients treated with PD-1 or PD-L1 inhibitors, CDK 4/6 inhibitors, or other immune-based therapy are eligible.

Exclusion Criteria:

* T4 tumors including inflammatory breast cancer
* Patients with distant metastatic disease
* Lumpectomy performed prior to study entry
* Patients with any history of prior radiation therapy in the affected breast
* Patients with a prior history of ipsilateral invasive breast cancer; (patients with previous ipsilateral/contralateral DCIS or previous contralateral invasive breast cancer treated with anti-cancer therapy are eligible)
* Patients with invasive lobular carcinoma
* Patients who have multicentric disease
* Patients treated with neoadjuvant hormonal therapy only are not eligible
* Patients who are medically unfit to undergo surgical resection
* Patients without breast biopsy marker documented by imaging at tumor bed site prior to initiation of neoadjuvant therapy
* Patients with one or more of the following imaging criteria from any of the 3 imaging modalities after completion of NCT demonstrating incomplete radiologic response are not eligible:

  * Mammogram with malignant appearing calcifications or mass > 1 cm; or
  * Ultrasound with a hypoechoic area > 2 cm; or
  * Breast MRI demonstrating a residual mass with rapid rise and washout type III kinetics.
* Psychiatric or addictive disorders or other conditions that, in the opinion of the investigator, would preclude the patient from meeting the study requirements or interfere with interpretation of study results
* Pregnancy or lactation at the time of study registration; (Note: Pregnancy testing according to institutional standards for women of childbearing potential must be performed within 2 weeks prior to study registration.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2017-04-13 (Actual); Primary Completion 2019-07-05 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with pCR | Up to 18 months
  The proportion of tumor bed biopsies that are negative among those who are shown to have pCR at surgery will be determined. The point estimate and 95% confidence interval will be calculated.

SECONDARY OUTCOMES:
Improvement of negative predictive value | Up to 18 months
  Analysis will be performed to assess the improvement in the negative predictive value of the trimodality imaging algorithm when the results of tumor bed biopsy are added.
Incidence of adverse events associated with tumor bed biopsy | Up to 18 months
  Descriptive analysis will be performed to determine the frequencies of adverse events associated with tumor bed biopsy.
Number of needle cores performed | Up to 18 months
  Descriptive analysis will be performed to determine the distribution of the number of needle cores performed and the proportion of clips retrieved.
Proportion of clips retrieved | Up to 18 months
  Descriptive analysis will be performed.
Residual cancer burden score | Up to 18 months
  Descriptive analysis will be performed to determine the distribution of residual cancer burden score.
Trimodality imaging algorithm +/- biopsy as a predictor of pCR | Up to18 months
  Analysis will be performed to assess the improvement in the negative predictive value of the trimodality imaging algorithm when the results of tumor bed biopsy are added.

OTHER OUTCOMES:
Molecular makers from tumor and blood samples | Up to 18 months
  Analysis to assess the association of molecular markers with response to neoadjuvant therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Basik, Principal Investigator — NRG Oncology
Locations (381):
- United States (377):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - University of South Alabama Mitchell Cancer Institute, Mobile, Alabama
  - Cancer Center at Saint Joseph's, Phoenix, Arizona
  - Banner University Medical Center - Tucson, Tucson, Arizona
  - University of Arizona Cancer Center-North Campus, Tucson, Arizona
  - Mercy Hospital Fort Smith, Fort Smith, Arkansas
  - Kaiser Permanente-Deer Valley Medical Center, Antioch, California
  - Sutter Auburn Faith Hospital, Auburn, California
  - Sutter Cancer Centers Radiation Oncology Services-Auburn, Auburn, California
  - Alta Bates Summit Medical Center-Herrick Campus, Berkeley, California
  - Mills-Peninsula Medical Center, Burlingame, California
  - Sutter Cancer Centers Radiation Oncology Services-Cameron Park, Cameron Park, California
  - Eden Hospital Medical Center, Castro Valley, California
  - Sutter Davis Hospital, Davis, California
  - Epic Care-Dublin, Dublin, California
  - Bay Area Breast Surgeons Inc, Emeryville, California
  - Epic Care Partners in Cancer Care, Emeryville, California
  - Kaiser Permanente-Fremont, Fremont, California
  - Palo Alto Medical Foundation-Fremont, Fremont, California
  - Fresno Cancer Center, Fresno, California
  - Kaiser Permanente-Fresno, Fresno, California
  - Los Angeles County-USC Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - Contra Costa Regional Medical Center, Martinez, California
  - Memorial Medical Center, Modesto, California
  - Kaiser Permanente-Modesto, Modesto, California
  - Palo Alto Medical Foundation-Camino Division, Mountain View, California
  - Palo Alto Medical Foundation-Gynecologic Oncology, Mountain View, California
  - Sutter Cancer Research Consortium, Novato, California
  - Alta Bates Summit Medical Center - Summit Campus, Oakland, California
  - Bay Area Tumor Institute, Oakland, California
  - Kaiser Permanente Oakland-Broadway, Oakland, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Palo Alto Medical Foundation Health Care, Palo Alto, California
  - Stanford Cancer Institute Palo Alto, Palo Alto, California
  - Keck Medical Center of USC Pasadena, Pasadena, California
  - Kaiser Permanente-Rancho Cordova Cancer Center, Rancho Cordova, California
  - Kaiser Permanente-Redwood City, Redwood City, California
  - Kaiser Permanente-Richmond, Richmond, California
  - Rohnert Park Cancer Center, Rohnert Park, California
  - Kaiser Permanente-Roseville, Roseville, California
  - Sutter Cancer Centers Radiation Oncology Services-Roseville, Roseville, California
  - Sutter Roseville Medical Center, Roseville, California
  - The Permanente Medical Group-Roseville Radiation Oncology, Roseville, California
  - Kaiser Permanente Downtown Commons, Sacramento, California
  - Sutter Medical Center Sacramento, Sacramento, California
  - Kaiser Permanente-South Sacramento, Sacramento, California
  - South Sacramento Cancer Center, Sacramento, California
  - Kaiser Permanente - Sacramento, Sacramento, California
  - Naval Medical Center -San Diego, San Diego, California
  - California Pacific Medical Center-Pacific Campus, San Francisco, California
  - Kaiser Permanente-San Francisco, San Francisco, California
  - Kaiser Permanente-Santa Teresa-San Jose, San Jose, California
  - Kaiser Permanente San Leandro, San Leandro, California
  - Kaiser Permanente-San Rafael, San Rafael, California
  - Kaiser San Rafael-Gallinas, San Rafael, California
  - Kaiser Permanente Medical Center - Santa Clara, Santa Clara, California
  - Palo Alto Medical Foundation-Santa Cruz, Santa Cruz, California
  - Kaiser Permanente-Santa Rosa, Santa Rosa, California
  - Sutter Pacific Medical Foundation, Santa Rosa, California
  - Kaiser Permanente Cancer Treatment Center, South San Francisco, California
  - Kaiser Permanente-South San Francisco, South San Francisco, California
  - Kaiser Permanente-Stockton, Stockton, California
  - Palo Alto Medical Foundation-Sunnyvale, Sunnyvale, California
  - Sutter Cancer Centers Radiation Oncology Services-Vacaville, Vacaville, California
  - Kaiser Permanente Medical Center-Vacaville, Vacaville, California
  - Kaiser Permanente-Vallejo, Vallejo, California
  - Sutter Solano Medical Center/Cancer Center, Vallejo, California
  - Kaiser Permanente-Walnut Creek, Walnut Creek, California
  - Epic Care Cyberknife Center, Walnut Creek, California
  - Rocky Mountain Cancer Centers-Aurora, Aurora, Colorado
  - University of Colorado Hospital, Aurora, Colorado
  - Boulder Community Hospital, Boulder, Colorado
  - Rocky Mountain Cancer Centers-Boulder, Boulder, Colorado
  - Denver Health Medical Center, Denver, Colorado
  - National Jewish Health-Main Campus, Denver, Colorado
  - The Women's Imaging Center, Denver, Colorado
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Presbyterian - Saint Lukes Medical Center - Health One, Denver, Colorado
  - Rocky Mountain Cancer Centers-Midtown, Denver, Colorado
  - SCL Health Saint Joseph Hospital, Denver, Colorado
  - Rocky Mountain Cancer Centers-Rose, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - Western Surgical Care, Denver, Colorado
  - Mountain Blue Cancer Care Center - Swedish, Englewood, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - National Jewish Health-Western Hematology Oncology, Golden, Colorado
  - Saint Mary's Hospital and Regional Medical Center, Grand Junction, Colorado
  - Grand Valley Oncology, Grand Junction, Colorado
  - North Colorado Medical Center, Greeley, Colorado
  - Good Samaritan Medical Center, Lafayette, Colorado
  - Rocky Mountain Cancer Centers-Littleton, Littleton, Colorado
  - Rocky Mountain Cancer Centers-Sky Ridge, Lone Tree, Colorado
  - McKee Medical Center, Loveland, Colorado
  - National Jewish Health-Northern Hematology Oncology, Thornton, Colorado
  - SCL Health Lutheran Medical Center, Wheat Ridge, Colorado
  - Smilow Cancer Center/Yale-New Haven Hospital, New Haven, Connecticut
  - Yale University, New Haven, Connecticut
  - Beebe Medical Center, Lewes, Delaware
  - Delaware Clinical and Laboratory Physicians PA, Newark, Delaware
  - Helen F Graham Cancer Center, Newark, Delaware
  - Medical Oncology Hematology Consultants PA, Newark, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Beebe Health Campus, Rehoboth Beach, Delaware
  - TidalHealth Nanticoke / Allen Cancer Center, Seaford, Delaware
  - Christiana Care Health System-Wilmington Hospital, Wilmington, Delaware
  - John Fitzgerald Kennedy Medical Center, Atlantis, Florida
  - University of Florida Health Science Center - Gainesville, Gainesville, Florida
  - Memorial Regional Hospital/Joe DiMaggio Children's Hospital, Hollywood, Florida
  - Orlando Health Cancer Institute, Orlando, Florida
  - Memorial Hospital West, Pembroke Pines, Florida
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Piedmont Hospital, Atlanta, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Emory Saint Joseph's Hospital, Atlanta, Georgia
  - Dekalb Medical Center, Decatur, Georgia
  - Piedmont Fayette Hospital, Fayetteville, Georgia
  - Medical Center of Central Georgia, Macon, Georgia
  - Hawaii Cancer Care Inc - Waterfront Plaza, Honolulu, Hawaii
  - Island Urology, Honolulu, Hawaii
  - Queen's Cancer Cenrer - POB I, Honolulu, Hawaii
  - Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Hawaii Cancer Care Inc-Liliha, Honolulu, Hawaii
  - Kuakini Medical Center, Honolulu, Hawaii
  - Queen's Cancer Center - Kuakini, Honolulu, Hawaii
  - The Cancer Center of Hawaii-Liliha, Honolulu, Hawaii
  - Kaiser Permanente Moanalua Medical Center, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Wilcox Memorial Hospital and Kauai Medical Clinic, Lihue, Hawaii
  - Hawaii Cancer Care - Westridge, ‘Aiea, Hawaii
  - Pali Momi Medical Center, ‘Aiea, Hawaii
  - Queen's Cancer Center - Pearlridge, ‘Aiea, Hawaii
  - The Cancer Center of Hawaii-Pali Momi, ‘Aiea, Hawaii
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Alphonsus Cancer Care Center-Caldwell, Caldwell, Idaho
  - Kootenai Health - Coeur d'Alene, Coeur d'Alene, Idaho
  - Walter Knox Memorial Hospital, Emmett, Idaho
  - Idaho Urologic Institute-Meridian, Meridian, Idaho
  - Saint Alphonsus Cancer Care Center-Nampa, Nampa, Idaho
  - Kootenai Clinic Cancer Services - Post Falls, Post Falls, Idaho
  - Kootenai Cancer Clinic, Sandpoint, Idaho
  - Rush - Copley Medical Center, Aurora, Illinois
  - Northwestern University, Chicago, Illinois
  - John H Stroger Jr Hospital of Cook County, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Carle at The Riverfront, Danville, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Northwestern Medicine Lake Forest Hospital, Lake Forest, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Marjorie Weinberg Cancer Center at Loyola-Gottlieb, Melrose Park, Illinois
  - Trinity Medical Center, Moline, Illinois
  - Good Samaritan Regional Health Center, Mount Vernon, Illinois
  - UC Comprehensive Cancer Center at Silver Cross, New Lenox, Illinois
  - University of Chicago Medicine-Orland Park, Orland Park, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - The Carle Foundation Hospital, Urbana, Illinois
  - Rush-Copley Healthcare Center, Yorkville, Illinois
  - Deaconess Clinic Downtown, Evansville, Indiana
  - Parkview Hospital Randallia, Fort Wayne, Indiana
  - Parkview Regional Medical Center, Fort Wayne, Indiana
  - Goshen Center for Cancer Care, Goshen, Indiana
  - Chancellor Center for Oncology, Newburgh, Indiana
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - Coffeyville Regional Medical Center, Coffeyville, Kansas
  - Central Care Cancer Center - Garden City, Garden City, Kansas
  - Central Care Cancer Center - Great Bend, Great Bend, Kansas
  - HaysMed University of Kansas Health System, Hays, Kansas
  - University of Kansas Cancer Center, Kansas City, Kansas
  - Kansas Institute of Medicine Cancer and Blood Center, Lenexa, Kansas
  - Minimally Invasive Surgery Hospital, Lenexa, Kansas
  - Olathe Health Cancer Center, Olathe, Kansas
  - Menorah Medical Center, Overland Park, Kansas
  - University of Kansas Cancer Center-Overland Park, Overland Park, Kansas
  - University of Kansas Hospital-Indian Creek Campus, Overland Park, Kansas
  - Ascension Via Christi - Pittsburg, Pittsburg, Kansas
  - Salina Regional Health Center, Salina, Kansas
  - University of Kansas Health System Saint Francis Campus, Topeka, Kansas
  - University of Kansas Hospital-Westwood Cancer Center, Westwood, Kansas
  - Louisiana State University Health Science Center, New Orleans, Louisiana
  - University Medical Center New Orleans, New Orleans, Louisiana
  - Anne Arundel Medical Center, Annapolis, Maryland
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - UM Upper Chesapeake Medical Center, Bel Air, Maryland
  - Lahey Hospital and Medical Center, Burlington, Massachusetts
  - Winchester Hospital, Winchester, Massachusetts
  - Henry Ford Cancer Institute-Downriver, Brownstown, Michigan
  - Henry Ford Macomb Hospital-Clinton Township, Clinton Township, Michigan
  - Henry Ford Medical Center-Fairlane, Dearborn, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Allegiance Health, Jackson, Michigan
  - Henry Ford Medical Center-Columbus, Novi, Michigan
  - Henry Ford West Bloomfield Hospital, West Bloomfield, Michigan
  - Sanford Joe Lueken Cancer Center, Bemidji, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Cambridge Medical Center, Cambridge, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Fairview Clinics and Surgery Center Maple Grove, Maple Grove, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Health Partners Inc, Minneapolis, Minnesota
  - Monticello Cancer Center, Monticello, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - Fairview Lakes Medical Center, Wyoming, Minnesota
  - Saint Louis Cancer and Breast Institute-Ballwin, Ballwin, Missouri
  - Central Care Cancer Center - Bolivar, Bolivar, Missouri
  - Cox Cancer Center Branson, Branson, Missouri
  - Siteman Cancer Center at Saint Peters Hospital, City of Saint Peters, Missouri
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - Centerpoint Medical Center LLC, Independence, Missouri
  - Freeman Health System, Joplin, Missouri
  - Mercy Hospital Joplin, Joplin, Missouri
  - Truman Medical Centers, Kansas City, Missouri
  - The University of Kansas Cancer Center-South, Kansas City, Missouri
  - Research Medical Center, Kansas City, Missouri
  - University of Kansas Cancer Center - North, Kansas City, Missouri
  - University of Kansas Cancer Center - Lee's Summit, Lee's Summit, Missouri
  - Delbert Day Cancer Institute at PCRMC, Rolla, Missouri
  - Mercy Clinic-Rolla-Cancer and Hematology, Rolla, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Saint Louis Cancer and Breast Institute-South City, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Mercy Hospital South, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - Siteman Cancer Center at Christian Hospital, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Mercy Hospital Washington, Washington, Missouri
  - Community Hospital of Anaconda, Anaconda, Montana
  - Billings Clinic Cancer Center, Billings, Montana
  - Saint Vincent Healthcare, Billings, Montana
  - Saint Vincent Frontier Cancer Center, Billings, Montana
  - Bozeman Deaconess Hospital, Bozeman, Montana
  - Saint James Community Hospital and Cancer Treatment Center, Butte, Montana
  - Benefis Healthcare- Sletten Cancer Institute, Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Saint Peter's Community Hospital, Helena, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Community Medical Hospital, Missoula, Montana
  - The Cancer Institute of New Jersey Hamilton, Hamilton, New Jersey
  - Rutgers Cancer Institute of New Jersey-Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Roswell Park Cancer Institute, Buffalo, New York
  - Mount Sinai Union Square, New York, New York
  - Mount Sinai West, New York, New York
  - Mount Sinai Hospital, New York, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - SUNY Upstate Medical Center-Community Campus, Syracuse, New York
  - Montefiore Medical Center-Einstein Campus, The Bronx, New York
  - Montefiore Medical Center-Weiler Hospital, The Bronx, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Atrium Health Pineville/LCI-Pineville, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Wake Forest University at Elkin, Elkin, North Carolina
  - Wake Forest University at Lexington, Lexington, North Carolina
  - Atrium Health Union/LCI-Union, Monroe, North Carolina
  - Wake Forest University at Mount Airy, Mount Airy, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - UHHS-Chagrin Highlands Medical Center, Beachwood, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - UH Seidman Cancer Center at Saint John Medical Center, Westlake, Ohio
  - UHHS-Westlake Medical Center, Westlake, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Mercy Hospital Oklahoma City, Oklahoma City, Oklahoma
  - Saint Alphonsus Medical Center-Baker City, Baker City, Oregon
  - Saint Alphonsus Medical Center-Ontario, Ontario, Oregon
  - Jefferson Abington Hospital, Abington, Pennsylvania
  - UPMC-Heritage Valley Health System Beaver, Beaver, Pennsylvania
  - Christiana Care Health System-Concord Health Center, Chadds Ford, Pennsylvania
  - Ephrata Cancer Center, Ephrata, Pennsylvania
  - Ephrata Community Hospital, Ephrata, Pennsylvania
  - Adams Cancer Center, Gettysburg, Pennsylvania
  - UPMC Cancer Centers - Arnold Palmer Pavilion, Greensburg, Pennsylvania
  - Cherry Tree Cancer Center, Hanover, Pennsylvania
  - UPMC Pinnacle Harrisburg, Harrisburg, Pennsylvania
  - UPMC Pinnacle Cancer Center/Community Osteopathic Campus, Harrisburg, Pennsylvania
  - UPMC-Johnstown/John P. Murtha Regional Cancer Center, Johnstown, Pennsylvania
  - Sechler Family Cancer Center, Lebanon, Pennsylvania
  - UPMC Cancer Center at UPMC McKeesport, McKeesport, Pennsylvania
  - UPMC Hillman Cancer Center in Coraopolis, Moon Township, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - UPMC-Magee Womens Hospital, Pittsburgh, Pennsylvania
  - UPMC-Presbyterian Hospital, Pittsburgh, Pennsylvania
  - UPMC-Saint Margaret, Pittsburgh, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - UPMC-Shadyside Hospital, Pittsburgh, Pennsylvania
  - UPMC-Passavant Hospital, Pittsburgh, Pennsylvania
  - UPMC-Saint Clair Hospital Cancer Center, Pittsburgh, Pennsylvania
  - UPMC Cancer Center at UPMC Northwest, Seneca, Pennsylvania
  - UPMC Uniontown Hospital Radiation Oncology, Uniontown, Pennsylvania
  - UPMC Washington Hospital Radiation Oncology, Washington, Pennsylvania
  - Reading Hospital, West Reading, Pennsylvania
  - Wexford Health and Wellness Pavilion, Wexford, Pennsylvania
  - WellSpan Health-York Cancer Center, York, Pennsylvania
  - WellSpan Health-York Hospital, York, Pennsylvania
  - Women and Infants Hospital, Providence, Rhode Island
  - Prisma Health Cancer Institute - Spartanburg, Boiling Springs, South Carolina
  - Prisma Health Cancer Institute - Easley, Easley, South Carolina
  - Prisma Health Cancer Institute - Butternut, Greenville, South Carolina
  - Prisma Health Cancer Institute - Faris, Greenville, South Carolina
  - Prisma Health Greenville Memorial Hospital, Greenville, South Carolina
  - Prisma Health Cancer Institute - Eastside, Greenville, South Carolina
  - Prisma Health Cancer Institute - Greer, Greer, South Carolina
  - Prisma Health Cancer Institute - Seneca, Seneca, South Carolina
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Vanderbilt-Ingram Cancer Center Cool Springs, Franklin, Tennessee
  - Baptist Memorial Hospital and Cancer Center-Memphis, Memphis, Tennessee
  - Vanderbilt Breast Center at One Hundred Oaks, Nashville, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Houston Methodist Hospital, Houston, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - Doctor's Hospital of Laredo, Laredo, Texas
  - Scott and White Healthcare Round Rock, Round Rock, Texas
  - Houston Methodist Sugar Land Hospital, Sugar Land, Texas
  - Scott and White Memorial Hospital, Temple, Texas
  - Farmington Health Center, Farmington, Utah
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - South Jordan Health Center, South Jordan, Utah
  - Sentara Cancer Institute at Sentara CarePlex Hospital, Hampton, Virginia
  - Sentara Leigh Hospital, Norfolk, Virginia
  - Sentara Norfolk General Hospital, Norfolk, Virginia
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia
  - Sentara Virginia Beach General Hospital, Virginia Beach, Virginia
  - Sentara Princess Anne Hospital, Virginia Beach, Virginia
  - United Hospital Center, Bridgeport, West Virginia
  - WVUH-Berkely Medical Center, Martinsburg, West Virginia
  - West Virginia University Healthcare, Morgantown, West Virginia
  - Camden Clark Medical Center, Parkersburg, West Virginia
  - Aurora Cancer Care-Southern Lakes VLCC, Burlington, Wisconsin
  - Aurora Health Center-Fond du Lac, Fond du Lac, Wisconsin
  - Aurora Health Care Germantown Health Center, Germantown, Wisconsin
  - Aurora Cancer Care-Grafton, Grafton, Wisconsin
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - Aurora Cancer Care-Kenosha South, Kenosha, Wisconsin
  - Aurora Bay Area Medical Group-Marinette, Marinette, Wisconsin
  - Aurora Cancer Care-Milwaukee, Milwaukee, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Aurora Sinai Medical Center, Milwaukee, Wisconsin
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin
  - Vince Lombardi Cancer Clinic - Oshkosh, Oshkosh, Wisconsin
  - Aurora Cancer Care-Racine, Racine, Wisconsin
  - Vince Lombardi Cancer Clinic-Sheboygan, Sheboygan, Wisconsin
  - Aurora Medical Center in Summit, Summit, Wisconsin
  - Vince Lombardi Cancer Clinic-Two Rivers, Two Rivers, Wisconsin
  - Aurora Cancer Care-Milwaukee West, Wauwatosa, Wisconsin
  - Aurora West Allis Medical Center, West Allis, Wisconsin
  - Cheyenne Regional Medical Center-West, Cheyenne, Wyoming
  - Billings Clinic-Cody, Cody, Wyoming
  - Welch Cancer Center, Sheridan, Wyoming
- Canada (4):
  - University Health Network-Princess Margaret Hospital, Toronto, Ontario
  - CHUM - Centre Hospitalier de l'Universite de Montreal, Montreal, Quebec
  - The Research Institute of the McGill University Health Centre (MUHC), Montreal, Quebec
  - Jewish General Hospital, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Basik M, Cecchini RS, De Los Santos JF, Umphrey HR, Julian TB, Mamounas EP, White JR, Lucas PC, Balanoff CR, Tan AR, Weber JJ, Edmonson DA, Brown-Glaberman UA, Diego EJ, Teshome M, Matsen CB, Seaward SA, Wapnir IL, Wagner JL, Tjoe JA, Thompson AM, Wolmark N. Breast Tumor-Bed Biopsy for Pathological Complete Response Prediction: The NRG-BR005 Nonrandomized Clinical Trial. JAMA Surg. 2025 Jul 1;160(7):723-731. doi: 10.1001/jamasurg.2025.1072. PMID 40332918
- [Derived] Gharzai LA, Szczygiel LA, Shumway DA, Bandos H, Julian TB, Mamounas EP, White J, De Los Santos JF, Basik M, Ganz PA, Jagsi R. A qualitative study to evaluate physician attitudes regarding omission of surgery among exceptional responders to neoadjuvant systemic therapy for breast cancer (NRG-CC006). Breast Cancer Res Treat. 2021 Jun;187(3):777-784. doi: 10.1007/s10549-021-06172-0. Epub 2021 Mar 19. PMID 33740205